CLINICAL TRIAL: NCT05026996
Title: A Single-dose, Open-label, Parallel-group Study to Assess the Pharmacokinetics of Pelacarsen (TQJ230) in Participants With Mild Hepatic Impairment Compared to Matched Healthy Participants
Brief Title: Study to Assess the Pharmacokinetics of Pelacarsen (TQJ230) in Participants With Mild Hepatic Impairment Compared to Matched Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTQJ230A12202
Record Dates: First submitted 2021-08-04; First posted 2021-08-30 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hepatic Impairment
Keywords: CTQJ230; Hepatic Impairment; Subcutaneous injection; single-dose
MeSH Terms: interventions — pelacarsen

STUDY DESIGN:
Intervention Model Description: This was a Phase I, open-label, single dose, parallel-group study in participants with mild HI (n=8) and matched healthy participants with normal hepatic function (n=8) designed to evaluate the PK of pelacarsen. Participants were matched by gender, age (± 10 years), and body weight (± 15%).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mild hepatic impairment patients (Experimental): Participants with mild hepatic impairment
  Interventions: Drug: Pelacarsen
- Healthy participants (Experimental): Matched healthy participants with normal hepatic function
  Interventions: Drug: Pelacarsen

INTERVENTIONS:
Drug: Pelacarsen — Single subcutaneous injection of pelacarsen
  Other Names: TQJ230

SUMMARY:
This was a Phase I, open-label, single-dose, parallel-group study in participants with mild hepatic impairment (HI) and healthy matched control participants with normal hepatic function designed to evaluate the PK of pelacarsen following a single 80 mg s.c. dose. Participants were matched by gender, age (±10 years), and body weight (±15%).

DETAILED DESCRIPTION:
The study consisted of a Screening period of up to 28 days, followed by Baseline evaluations on Day -1. Participants who met the eligibility criteria at Screening were admitted to Baseline evaluations.

On Day 1, participants received a single s.c. injection of 80 mg pelacarsen followed by PK sampling up to Day 60 (±3 days). Participants were domiciled for at least 4 overnight stays (Day -1 through Day 4) for PK sample collection up to 72 hours postdose and were to return to the study site on 3 occasions (Days 8, 30 [±2 days], and 60 [±3 days]) for additional PK sample collection.

Study Completion evaluation occurred with the completion of Day 60 (±3 days) assessments. The total study duration for each participant was expected to be up to a maximum of 89 (±3) days, including the Screening period.

A post study safety contact took place on Day 112, approximately 16 weeks after dosing.

ELIGIBILITY:
Inclusion Criteria:

All participants

1. Signed informed consent must be obtained prior to participation in the study.
2. Male and non-child bearing potential female participants, 18 to 75 years of age (inclusive), at Screening.
3. Participants must weigh at least 50 kg to participate in the study, and must have a BMI within the range of 18.0 - 38.0 kg/m2, at Screening.
4. Ability to communicate well with the investigator, to understand and comply with the requirements of the study.
5. Must be a non-smoker or agree to smoke no more than 5 cigarettes (or equivalent) per day from Screening until Study Completion.

   Participants with mild HI (Group 2)
6. Participants must have a prior diagnosis of liver cirrhosis and mild HI as defined by the Child Pugh classification with a score of 5-6, inclusive (Class A)
7. Participants have been clinically stable and had no worsening of more than 1 point in Child Pugh score within 1 month prior to dosing of study treatment.
8. Seated vital signs must be within the following ranges at Screening and Baseline:

   * Body temperature between 35.0 to 37.5°C, inclusive;
   * Systolic blood pressure between 100 to 159 mmHg, inclusive;
   * Diastolic blood pressure between 60 to 109 mmHg, inclusive;
   * Pulse rate between 45 - 99 bpm, inclusive.
9. Participants with other stable medical disorders such as controlled diabetes, hyperlipidemia, hypothyroidism, etc., may be eligible as long as they are considered appropriate for enrollment as determined by the investigator by medical history, physical examination, ECG, and clinical laboratory tests at Screening.

   Healthy control participants (Group 1)
10. Each participant must match 1:1 in gender, age (± 10 years), and body weight (± 15%) to a participant with mild HI.
11. Seated vital signs must be within the following ranges at Screening and Baseline:

    * Body temperature between 35.0 to 37.5°C, inclusive;
    * Systolic blood pressure between 89 to 139 mmHg, inclusive;
    * Diastolic blood pressure between 50 to 89 mmHg, inclusive;
    * Pulse rate between 45 to 90 bpm, inclusive.
12. Participants must be in good health as determined by medical history, physical examination, ECG, and clinical laboratory tests at Screening.

Exclusion Criteria:

All participants

1. Use of other investigational drugs within 5 half-lives or 30 days prior to dosing of study treatment, whichever is longer.
2. History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes.
3. Treatment with any oligonucleotide (with an exception for COVID 19 vaccines) or SiRNA within 9 months prior to Screening.
4. Participants who received any COVID 19 vaccination and/or have not completed their full COVID-19 vaccination regimen within 14 days prior to Screening.
5. Women of child bearing potential, defined as all women physiologically capable of becoming pregnant. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least 6 weeks prior to the first dosing. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential.
6. Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 16 weeks after stopping study treatment. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, male participants must not donate sperm for the time period specified above.
7. Known history of, or current clinically significant arrhythmias, history of prolonged QT interval corrected by Fridericia's formula (QTcF), QTcF > 450 msec (males), or QTcF > 460 msec (females) at Screening.
8. History of immunodeficiency diseases or have a positive HIV test result at Screening.
9. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years of Screening, regardless of whether there is evidence of local recurrence or metastases.
10. Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing of study treatment.
11. Platelet count ≤ LLN at Screening or Baseline.
12. History of unhealthy alcohol use within 12 months prior to dosing of study treatment, as defined by a recurring pattern of either binge drinking (≥ 5 drinks over 2 3 hours on ≥ 5 days/month) or heavy drinking (≥ 8 drinks/week in females or > 15 drinks/week in males). A "drink" definition includes: 12 ounces of 5% beer, 8 ounces of 7% malt liquor, 5 ounces of 12% wine or 1.5 ounces of 40% spirits.
13. Positive alcohol screen at Screening or Baseline.
14. History of drug abuse within the last 12 months or evidence of such abuse as indicated by the laboratory assay conducted during Screening or Baseline, unless the positive drug screen is due to prescription drug use that is approved by the investigator and Novartis.
15. Clinically significant illness (other than HI for participants in Group 2) within 2 weeks prior to dosing of study treatment that may jeopardize safety of the participant and/or alter the study results as judged by the investigator.
16. Significant glomerular disease (including but not limited to IgA nephropathy, diabetic nephropathy, systemic lupus erythematosus, etc.) with urinary protein-creatinine ratio > 500 mg/g (56.6 mg/mmol).
17. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs (apart from cholecystectomy), or which may jeopardize the participants in case of participation in the study. The investigator should make this determination in consideration of the participant's medical history.
18. Have tattoo(s) or scarring at or near the site of injection or any other condition which may interfere with injection site examination, in the opinion of the investigator.
19. Unwillingness or inability (e.g. physical or cognitive) to comply with study procedures, study treatment administration (i.e. injection), or schedule.

    Participants with mild HI (Group 2)
20. Presence of any non controlled and clinically significant disease that could affect the study outcome or that would place the participant at undue risk.
21. Severe complications of liver disease within the preceding 3 months of Screening.
22. Have received liver transplant at any time in the past.
23. Participants requiring paracentesis more than every 30 days for the management of ascites. Participants who are receiving diuretics to manage ascites may be enrolled and will be assigned the Child Pugh score for the degree of ascites while on diuretic treatment. The diuretic dose must have been stable for at least 14 days prior to dosing of study treatment.
24. Have transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.
25. Have acute hepatitis B or C infection at Screening or active infection requiring therapy that will not be completed before Screening.
26. Presence of moderate to severe impaired renal function as indicated by estimated glomerular filtration rate < 45 mL/min/1.73 m2 based on MDRD calculation.
27. Hemoglobin levels below 10.0 g/dL at Screening or Baseline.
28. Have encephalopathy Grade 3 or worse within 28 days prior to dosing of study treatment.
29. Have primary biliary cholangitis or biliary obstruction.
30. History of gastrointestinal bleeding within the past 3 months prior to Screening.
31. Clinically significant abnormal findings in physical examination or clinical laboratory evaluations not consistent with known liver disease.

    Healthy control participants (Group 1)
32. Any single parameter of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl-transferase (GGT), or alkaline phosphatase (ALP) exceeding 1.2 x upper limit of normal (ULN), total bilirubin ≥ 1.5 x ULN, or any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or total bilirubin at Screening or Baseline.
33. Hemoglobin levels more than 10% below LLN at Screening or Baseline.
34. Participants known to have Gilbert's syndrome.
35. Chronic hepatitis B or hepatitis C infection. A positive HBsAg test, or if standard local practice, a positive hepatitis B virus core antigen test, is an exclusion. Participants with a positive hepatitis C virus (HCV) antibodies (Ab) test should have HCV ribonucleic acid (RNA) levels measured. Participants with positive (detectable) HCV RNA should be excluded.
36. Are taking medications prohibited with the study treatment (see Section 6.2.2 for additional details on prohibited medication) or herbal supplements, prescribed medicinal use of cannabis/marijuana, within 14 days prior to dosing of study treatment.
37. Impaired renal function as indicated by clinically significantly abnormal creatinine or blood urea nitrogen and/or urea values, or abnormal urinary constituents at screening and/or baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of pelacarsen: Cmax | Day 1 (0 hour (pre-dose) 0.5 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour), Day 2, Day 3, Day 4, Day 8, Day 30 and Day 60
  The maximum (peak) observed drug concentration in after single-dose administration (mass x volume-1).
  To assess the PK properties of plasma pelacarsen after a single s.c. injection in participants with mild HI (Child-Pugh classification) as compared to matched healthy participants with normal hepatic function.
Pharmacokinetic parameters of pelacarsen: AUClast | Day 1 (0 hour (pre-dose) 0.5 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour), Day 2, Day 3, Day 4, Day 8, Day 30 and Day 60
  The area under the concentration-time curve (AUC) from time zero to the last measurable concentration sampling time (mass x time x volume-1).
  To assess the PK properties of plasma pelacarsen after a single s.c. injection in participants with mild HI (Child-Pugh classification) as compared to matched healthy participants with normal hepatic function.
Pharmacokinetic parameters of pelacarsen: AUCinf | Day 1 (0 hour (pre-dose) 0.5 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour), Day 2, Day 3, Day 4, Day 8, Day 30 and Day 60
  The AUC from time zero to infinity (mass x time x volume-1). To assess the PK properties of plasma pelacarsen after a single s.c. injection in participants with mild HI (Child-Pugh classification) as compared to matched healthy participants with normal hepatic function.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milosavljevic MN, Stefanovic SM, Pejcic AV. Potential Novel RNA-Targeting Agents for Effective Lipoprotein(a) Lowering: A Systematic Assessment of the Evidence From Completed and Ongoing Developmental Clinical Trials. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):1-12. doi: 10.1097/FJC.0000000000001429. PMID 37070852
- See also: Results for CTQJ230A12202 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18105
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1835